CLINICAL TRIAL: NCT04921813
Title: Investigation of the Efficiency of Three Dimensional Scoliosis Exercises and Balance-Coordination Exercises in the Conservative Treatment of Adolescent Idiopathic Scoliosis Patients.
Brief Title: Investigation of Conservative Treatment on Adolescent Idiopathic Scoliosis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, assistant professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BandırmaOnyediEylulU
Record Dates: First submitted 2021-02-07; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: rondomized controlled trail
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Schroth method + brace (Experimental): 3-dimensional scoliosis exercise program according to Schroth method + brace.
  Interventions: Other: 3 dimensional scoliosis exercise; Other: Brace treatment
- Schroth + balance-coordination exercises + brace. (Experimental): 3-dimensional scoliosis exercise program according to Schroth + balance-coordination exercises + brace.
  Interventions: Other: 3 dimensional scoliosis exercise; Other: Balance Exercise; Other: Brace treatment
- Brace (Experimental): Only brace treatment.
  Interventions: Other: Brace treatment
- healthy individuals (No Intervention): Age-matched control group

INTERVENTIONS:
Other: 3 dimensional scoliosis exercise — Schroth exercises
  Arms: Schroth + balance-coordination exercises + brace.; Schroth method + brace
Other: Balance Exercise — Balance-coordination exercises
  Arms: Schroth + balance-coordination exercises + brace.
Other: Brace treatment — Brace usage
  Arms: Brace; Schroth + balance-coordination exercises + brace.; Schroth method + brace

SUMMARY:
Aim: It was aimed to investigate the effectiveness of three-dimensional scoliosis exercises and balance-coordination exercises in patients with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Method: Thirty patients who were diagnosed with adolescent idiopathic scoliosis were randomly divided into three groups. The first group was treated with 3-dimensional scoliosis exercise program according to Schroth method, second group was treated with Schroth exercises and balance-coordination exercises in addition to brace. Exercises were performed for a total of 6 weeks (18 sessions). The third group was treated only with brace and the control group consisted of healthy individuals. Patients were assessed for their curve angle (Cobb method), rotation angle (scoliometer), spinal flexibility (anterior and lateral bending tests), quality of life (Scoliosis Research Society-22), cosmetic effects (Walter Reed Visual Rating Scale), balance parameters (Balance Master System NeuroCom International Inc. Clackamas, OR, USA ver 8.1), vertical perception (Subjective Vertical Detection test) and brain responses (electroencephalography) were assessed before and after treatment. SPSS 20.0 statistical program was used for data analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with adolescent idiopathic scoliosis between the ages of 10-16 and being deemed appropriate for brace use,
* Cobb angle between 20º -50º,
* To be able to continue the program to be applied,
* Not having a chronic disease that requires the use of any neurological or psychiatric medication, Hearing test results are within normal values,
* Parents allow the child to participate in the study

Exclusion Criteria:

* The patient has any contraindications to exercise,
* Previous spine surgery,
* Having a curvature of thoracic apex 6 or more,
* Having any mental problems,
* Scoliosis is not idiopathic but has occurred for different reasons (neurological, congenital, etc.),
* Presence of neurological, psychiatric, muscular, rheumatic or orthopedic diseases.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Balance and postural control parameters -Weight Bearing/Squat | Change from baseline balance and postural control parameters at 6 weeks, Change from baseline balance and postural control parameters at 1 year, Change from 6th weeks balance and postural control parameters at 1 year
  Weight Bearing/Squat (percentage, %): Weight bearing percentages of the right and left feet were measured at 0°, 30°, 60°, 90° knee flexion.
Cobb Angle | Change from baseline Cobb angle at 1 year
  Cobb Angle (degree): The degree of curvature in the coronal plane is measured radiographically according to the Cobb method
Angle of Trunk Rotation | Change from baseline Angle of Trunk Rotation at 6 weeks, Change from baseline Angle of Trunk Rotation at 1 year, Change from 6th weeks Angle of Trunk Rotation at 1 year
  ATR - Angle of Trunk Rotation (degree): Measurement of trunk rotation angle/degree is the most appropriate method used in the clinical evaluation of scoliosis.
Evaluation of subjective visual vertical perception | Change from baseline subjective visual vertical perception at 6 weeks, Change from baseline subjective visual vertical perception at 1 year, Change from 6th weeks subjective visual vertical perception at 1 year
  Evaluation of subjective visual vertical perception (degree): Subjects were asked to manually verticalize the deviated laser line projected on a wall 1 m away in a room that is dark enough to prevent them from taking visual references while standing. Photographs were recorded during this process.
Electroencephalography (EEG) | Change from baseline EEG at 6 weeks
  In EEG recordings, epochs of 1000 ms before and 1000 ms after the stimulus were created. In these sweeps, those with amplitudes greater than ±50 μV in the EOG electrode channels and those with noise were removed. The files obtained for each individual were baseline corrected and filtered with a digital bandpass filter with 0.5 - 48 Hz limit values (12 dB/oct and zero phase shift, Neuroscan 4.5 ). After the filtering process, the mean (average) file was created for each individual.
  In measuring the amplitudes of the electrophysiological responses, the responses with the largest amplitudes between 0-1000 ms were measured and evaluated in µV. EEG recordings were taken from 64 channels. However, PO3, POZ and PO4 electrodes in the parieto-occipital region were investigated as these are the primary areas for visual stimuli.
The Dicotic Listening Paradigm: | Change from baseline The Dicotic Listening Paradigm parameters at 6 weeks
  There are 30 different (heteronymous) and 6 identical (homonymous) combinations for syllables. It was applied at 78.9 dB SPL (sound pressure level) in dichotic application. . Three rounds, with an average session duration of 7.5 minutes, and a total of approximately 25-30 minutes of test with intervals. In the dichotic application, the participants were first asked to respond without paying attention to any of their ears (non-forced/NF). In the following session, the participants were told to direct their attention to their right ear (forced right ear attention/FR) and to direct their attention to their left ear (forced left ear attention/FL).
Assessment of health-related quality of life | Change from baseline The Scoliosis Research Society - 22 questionnaire at 6 weeks, Change from baseline The Scoliosis Research Society - 22 questionnaire at 1 year, Change from 6th weeks The Scoliosis Research Society - 22 questionnaire at 1 year
  The Scoliosis Research Society - 22 questionnaire (SRS-22) is a health-related quality of life questionnaire designed specifically for patients with spinal deformities. SRS-22 consists of the sub-headings of function, pain, body image, mental health and satisfaction with treatment and includes 22 questions in total.
Balance and postural control parameters-Modified Clinical test of Sensory Interaction on Balance | Change from baseline balance and postural control parameters at 6 weeks, Change from baseline balance and postural control parameters at 1 year, Change from 6th weeks balance and postural control parameters at 1 year
  Modified Clinical test of Sensory Interaction on Balance (degrees per second,°/sn): Body center of gravity is expressed as the ratio of swing speed and distance to time. Body center of gravity is the ratio between distance traveled (expressed in degrees) and trial time (10 sn).
  Average body center of gravity swing rate (degrees per second) i) Eyes open on hard ground, ii) Eyes closed on hard ground, iii) On soft ground, eyes open and iv) It was measured in four different situations with eyes closed on soft ground.
Balance and postural control parameters-Limit of stability | Change from baseline balance and postural control parameters at 6 weeks, Change from baseline balance and postural control parameters at 1 year, Change from 6th weeks balance and postural control parameters at 1 year
  Limit of stability (% and °/sn): It is used to determine the limits of body stability. Reaction time (sec), movement speed (degrees / sec), end point reached (%), maximum end point (%) in 8 directions: front, right front, right, right back, rear, left back, left, left front and measurements were taken in terms of directional control (%).

IPD SHARING:
Plan to Share IPD: No